CLINICAL TRIAL: NCT04655378
Title: Recherche d'un Marqueur Pronostique de l'Atteinte rénale du Purpura Rhumatoïde de l'Enfant. Validation de la méthode de détection Des IgA1 Avec Gradient de la Glycosylation Par spectrométrie de Masse
Brief Title: Validation of the IgA1 Detection Method With Gradient Glycosylation by Mass Spectrometry as a Potential Marker of Renal Involvement in Pediatric Rheumatoid Purpura
Acronym: FOXIGA-2020
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2020-1/TAT-01
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Rheumatoid Purpura; Pediatric ALL
MeSH Terms: conditions — IgA Vasculitis; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples already in existence
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute Rheumatoid Purpura
  Interventions: Other: Mass Sepctrometry
- Rheumatoid Purpura in Remission
  Interventions: Other: Mass Sepctrometry
- Controls: Without infection, inflammatory or auto-immune pathology
  Interventions: Other: Mass Sepctrometry

INTERVENTIONS:
Other: Mass Sepctrometry — Mass spectrometry (LC/MS) of purified immunoglobulins

SUMMARY:
In this ancillary study on the FoxTreg cohort, the study investigators will select variables to input and thus develop two models (Linear Discriminant Analysis and Decision Tree). The aim of this study is to validate the method in terms of repeatability, reproducibility, control of pre-analytical conditions and sample conservation, to complete the screening of IgA glycosylation in individuals of the FoxTreg cohort and to refine the glycopeptide signature to predict renal involvement.

ELIGIBILITY:
Inclusion Criteria:

Patient sera from biobank of the FoxTreg study (NCT02317133)

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This is an ancillary study on the patient biobank of the FoxTreg study (NCT02317133). All these patients had given their consent for blood sampling and the conservation of biological samples within the Biological Resources Center (CRB) of Nîmes. A total of 97 patients were recruited, forming three groups:
  * Group A (n = 30): patients with active Rheumatoid Purpura according to the criteria of EULAR / PRES / PRINTO 2010 [Ozen et al. 2010].
  * Group B (n = 30): patients in remission of Rheumatoid Purpura according to the criteria of EULAR / PRES / PRINTO 2010 [Ozen et al. 2010].
  * Group C (n = 37): age-matched control subjects free of infectious / inflammatory / autoimmune pathology.
  For this "FoxIgA-2020" study, only sera collected from these patients not analyzed in the "FoxIgA" study will be used.
  Thus 52 samples will be analyzed for the FoxIgA-2020 study:
  * 10 sera from group A
  * 14 sera from group B
  * 28 sera of group C
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Glycopeptide signature of serum from children with Rheumatoid Purpura | Day 0
  Mass spectrometry to identify the glycopeptides present and their level

SECONDARY OUTCOMES:
Repeatability of mass spectrometry in measuring glycopeptide signature | Day 0
  Mass spectrometry to identify the glycopeptides present and their level
Reproducibility of mass spectrometry in measuring glycopeptide signature | Day 0
  Mass spectrometry to identify the glycopeptides present and their level
Control of conservation of samples for measuring glycopeptide signature | Day 0
  Mass spectrometry to identify the glycopeptides present and their level
Glycopeptide signature of serum from all patients of the cohort | Day 0
  Mass spectrometry to identify the glycopeptides present and their level
Difference between a normally glycosylated IgA and an IgA with GalNac polymer in Rheumatoid Purpura patients with / without renal impairment versus controls | Day 0
  Mass spectrometry to identify the glycopeptides present and their level
Number of subjects with IgA glycosylation abnormalities in Rheumatoid Purpura patient population with renal impairment polymer in Rheumatoid Purpura patients with / without renal impairment versus controls | Day 0
  Mass spectrometry of IgA
Percentage of subjects with IgA glycosylation abnormalities in Rheumatoid Purpura patient population with renal impairment polymer in Rheumatoid Purpura patients with / without renal impairment versus controls | Day 0
  Mass spectrometry of IgA
Number of subjects with IgA glycosylation abnormalities in each group | Day 0
  Mass spectrometry of IgA
Percentage of subjects with IgA glycosylation abnormalities in each group | Day 0
  Mass spectrometry of IgA
Serum immunoglobulin levels in patients with acute Rheumatoid Purpura and in remission | Day 0
  Mass spectrometry of immunoglobulins IgA, IgM and IgG (g/L)
Quantification of blood cell lines in patients with acute Rheumatoid Purpura and in remission. | Day 0
  Blood cell lines, particularly Treg and Breg (number/mm3)
Serum cytokine levels in patients with acute Rheumatoid Purpura and in remission | Day 0
  pg/ml of TGF-β, IL-1, IL-6, TNF-α, IL-8, IL-10 and IL-17
Bacterial Translocation in patients with Rheumatoid Purpura | Day 0
  Plasma levels of 16S rDNA (copies/µl)
Plasma levels of LBP in patients with Rheumatoid Purpura | Day 0
  µg/ml
Plasma levels of CD14s in patients with Rheumatoid Purpura | Day 0
  µg/ml
Bacterial diversity in the gut microbiota in patients with Rheumatoid Purpura | Day 0
  Diversity Index

CONTACTS AND LOCATIONS:
Overall Officials: Tu Anh TRAN, Principal Investigator — CHU de Nimes
Locations (2):
- France (2):
  - CHRU de Montpellier, Montpellier
  - CHU de Nimes, Nîmes

REFERENCES:
- [Background] Ozen S, Pistorio A, Iusan SM, Bakkaloglu A, Herlin T, Brik R, Buoncompagni A, Lazar C, Bilge I, Uziel Y, Rigante D, Cantarini L, Hilario MO, Silva CA, Alegria M, Norambuena X, Belot A, Berkun Y, Estrella AI, Olivieri AN, Alpigiani MG, Rumba I, Sztajnbok F, Tambic-Bukovac L, Breda L, Al-Mayouf S, Mihaylova D, Chasnyk V, Sengler C, Klein-Gitelman M, Djeddi D, Nuno L, Pruunsild C, Brunner J, Kondi A, Pagava K, Pederzoli S, Martini A, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO). EULAR/PRINTO/PRES criteria for Henoch-Schonlein purpura, childhood polyarteritis nodosa, childhood Wegener granulomatosis and childhood Takayasu arteritis: Ankara 2008. Part II: Final classification criteria. Ann Rheum Dis. 2010 May;69(5):798-806. doi: 10.1136/ard.2009.116657. PMID 20413568